CLINICAL TRIAL: NCT01312441
Title: Sustainability of 25-hydroxyvitamin D Levels, Inflammatory Reduction, and Endothelial Dysfunction After Repletion With Ergocalciferol in CKD Stage 5D
Brief Title: Sustainability of Vitamin D Levels After Repletion With Ergocalciferol In Chronic Kidney Disease Stage 5D
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Albany College of Pharmacy and Health Sciences (Other)
Collaborators: VA Office of Research and Development (U.S. Federal Agency); Hortense & Louis Rubin Dialysis Center (Other); Satellite Healthcare (Other)
Responsible Party: Principal Investigator, Darius Mason, PI, Albany College of Pharmacy and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00741; 10-023 (Other: Albany College of Pharmacy and Health Sciences)
Record Dates: First submitted 2011-03-09; First posted 2011-03-10 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Vitamin D Deficiency; Renal Failure Chronic Requiring Hemodialysis
Keywords: Vitamin D; Ergocalciferol
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Ergocalciferols

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ergocalciferol (Experimental): Ergocalciferol 50,000 IU by mouth once weekly for 6 months
  Interventions: Drug: Ergocalciferol
- Placebo (Placebo Comparator): Placebo by mouth once weekly for 6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ergocalciferol — Ergocalciferol capsules 50,000 IU once weekly for 6 months
  Other Names: Drisdol
  Arms: Ergocalciferol
Drug: Placebo — Placebo by mouth once weekly for 6 months
  Arms: Placebo

SUMMARY:
The prevalence of vitamin D deficiency increases as kidney function declines. As a result, many hemodialysis patients often have low levels of vitamin D. Recent evidence has shown that vitamin D supplementation may improve many aspects of poor health such as heart disease and inflammatory markers. The objectives of this study are to determine how supplementing dialysis patients with ergocalciferol increases vitamin D levels, how long vitamin D levels can be maintained after a 6 month treatment course, and to examine the effect of ergocalciferol on biomarkers of inflammation and vascular health.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Activated vitamin D administration
* On chronic hemodialysis for ≥ 6 months
* Use of a synthetic biocompatible dialysis membrane
* 25-hydroxyvitamin D levels < 30 ng/mL
* Corrected serum calcium < 10.2 mg/dL
* Serum phosphate < 7 mg/dL
* Iron replete (Ferritin > 200 ng/mL and transferrin saturation > 20%)

Exclusion Criteria:

* Current participation in any other investigational drug trial
* Vitamin D deficiency due to a heredity disorder
* Liver disease or failure
* Current or past treatment with ergocalciferol or cholecalciferol ≥ 2000 IU per day (within the past 6 months)
* Treatment with calcimimetics or bisphosphonates within the last 3 months
* Treatment with anti-epileptics or other medications that can effect vitamin D metabolism
* Malnutrition (serum albumin < 2.5 mg/dL)
* Pregnancy, positive pregnancy test or breastfeeding
* Malignancy or other significant inflammatory disease
* HIV/AIDS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-01; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
The sustainability of 25-hydroxy-vitamin D levels after 6 months of vitamin D replenishment with ergocalciferol | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Darius L Mason, Pharm.D., Principal Investigator — Albany College of Pharmacy and Health Sciences; Roy Mathew, MD, Principal Investigator — Stratton Veteran Affairs Medical Center
Locations (4):
- United States (4):
  - Stratton VA Medical Center, Albany, New York
  - Hortense and Louis Rubin Dialysis Center, Clifton Park, New York
  - Hortense and Louis Rubin Dialysis Center, Saratoga Springs, New York
  - Hortense and Louis Rubin Dialysis Center, Troy, New York